CLINICAL TRIAL: NCT05099263
Title: The Vivaer Procedure for Treatment of the Septal Swell Bodies for Airway Obstruction - A Prospective Open-Label Multicenter Study (SWELL)
Brief Title: The Vivaer Procedure for Treatment of the Septal Swell Bodies (SWELL)
Acronym: SWELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP1125
Record Dates: First submitted 2021-10-11; First posted 2021-10-29 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Vivaer Procedure (Experimental): The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants will undergo bilateral treatment of the nasal airway in a single study procedure session. Each side of the nose will be treated as follows:
  • Two (2) to six (6) nonoverlapping applications of RF energy are performed at the SSB per nostril.
  The default treatment settings will be used for the study: temperature 60 C, power 4 watts, treatment time 18 seconds, and cooling time 12 seconds. No repeat ("touch up") procedures will be permitted after the initial procedure through the end of the study (36 months).
  Interventions: Device: Vivaer Arc Stylus

INTERVENTIONS:
Device: Vivaer Arc Stylus — The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants in this study will undergo bilateral treatment of the nasal airway in a single study session.

SUMMARY:
Post-market study to access the clinical use of the Vivaer Arc Stylus to treat Septal Swell Bodies (SSB).

DETAILED DESCRIPTION:
Prospective, Open-Label, Multicenter, Single Arm Study of the Aerin Medical Vivaer ARC Stylus to treat Septal Swell Bodies (SSB) to improve symptoms in adults diagnosed with nasal obstruction attributed to SSB.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 to 85 years (inclusively).
2. Seeking treatment for nasal obstruction and willing to undergo an office-based procedure.
3. Baseline NOSE score ≥ 55.
4. Presence of SSB hypertrophy limiting visualization of the middle turbinate (MT) by more than 50%.
5. Reduction in size of the SSB after application of topical decongestant on a cotton plug directly to the SSB region.
6. Improvement in the symptoms of nasal obstruction after SSB decongestion suggesting that the SSB may play a role in nasal obstruction.
7. Willing and able to withhold anticoagulant medications during the perioperative period (3-day window on either side).
8. Willing and able to provide informed consent.
9. Willing and able to comply with the participant-specific requirements outlined in the study protocol.

Exclusion Criteria:

1. Rhinoplasty, septoplasty, inferior turbinate (IT) reduction, or other surgical nasal procedures within the preceding 6 months.
2. Severe case of any of the following: septal deviation, turbinate hypertrophy, polyps, or ptotic nose tip believed to be the primary contributor to the participant's nasal obstruction symptoms and warranting surgical intervention.
3. Any adjunctive surgical nasal procedure planned on the same day or within 3 months after the Vivaer procedure.
4. Known or suspected allergies or contraindications for any general or local anesthetic agents.
5. Known or suspected to be pregnant or is lactating.
6. Participating in another clinical research study.
7. Other medical conditions which in the opinion of the investigator would predispose the participant to poor wound healing or increased surgical risk, or poor compliance with the requirements of the study.
8. Known or suspected regular use of oxymetazoline (Afrin) nasal decongestant or oral steroids.
9. For sites participating in the CT substudy only: Active sinus condition (eg, significant sinus diseases, infection or polyp formation) identified by CT.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2024-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anais Laborde, Study Director — Aerin Medical
Locations (9):
- United States (9):
  - Colorado Otolaryngology Associates LLC, Colorado Springs, Colorado
  - Chicago Nasal and Sinus Center, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - Mount Sinai, New York, New York
  - Madison ENT, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Vanderbilt Asthma, Sinus & Allergy Program, Nashville, Tennessee
  - Alamo ENT Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
No data collected will be shared with other researchers participating in the study.

REFERENCES:
- [Result] Pritikin J, Silvers S, Rosenbloom J, Davis B, Signore AD, Sedaghat AR, Tajudeen BA, Schmale I, Lyons J, Corey J, Chandra R. Temperature-controlled radiofrequency device treatment of septal swell bodies for nasal airway obstruction: An open-label, single arm multicenter study. Int Forum Allergy Rhinol. 2023 Oct;13(10):1915-1925. doi: 10.1002/alr.23156. Epub 2023 Mar 27. PMID 36908245
- [Result] Pritikin J, Silvers S, Rosenbloom J, Davis B, Del Signore A, Sedaghat AR, Tajudeen BA, Schmale I, Chandra RK. Twenty-Four-Month Outcomes Following Temperature-Controlled Radiofrequency Treatment for Septal Swell Body Hypertrophy: An Open-Label, Single-Arm Multicenter Study. Int Forum Allergy Rhinol. 2025 Jun;15(6):651-654. doi: 10.1002/alr.23541. Epub 2025 Feb 12. No abstract available. PMID 39936254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 9 academic medical centers and clinics between August 25, 2021 and April 28, 2022. The First Participant enrolled on September 14, 2021 and the last participant enrolled on April 28, 2022.
Pre-assignment Details: There was no wash out or run in for this study. A subset of study sites were selected to participate in a substudy of the use of CT imaging to assess changes in the SBB after treatment.
Groups:
- Vivaer Procedure: The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants will undergo bilateral treatment of the nasal airway in a single study procedure session. Each side of the nose will be treated as follows:
  • Two (2) to six (6) nonoverlapping applications of RF energy are performed at the SSB per nostril.
  The default treatment settings will be used for the study: temperature 60 C, power 4 watts, treatment time 18 seconds, and cooling time 12 seconds. No repeat ("touch up") procedures will be permitted after the initial procedure through the end of the study (36 months).
  Vivaer Arc Stylus: The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants in this study will undergo bilateral treatment of the nasal airway in a single study session.
Period: Overall Study
Arm/Group | Vivaer Procedure
Started | 70
3-Month | 68 (less 1-LTF, 1-Participation External Procedure)
6-Month | 65 (less 2-participation in external procedure and 1-PD pregnancy)
12-Month | 62 (less 1 LTF and 2 excluded due to participation in externalprocedure)
Completed (A total of 70 patients were treated and 62 reached (12M Visit) 1 year. The study is still in follow-up through 36M (3 years)) | 0
Not Completed | 70

BASELINE CHARACTERISTICS:
Groups:
- Single Arm - Vivaer Treatment: target population for this study is adults suffering from symptoms attributed to NAO with evidence of SSB obstruction of the airway which may or may not include hypertrophied turbinates. This study requires severe or extreme symptoms demonstrated by a NOSE Scale score ≥ 55 and determination by the investigator that the SSBs are the primary or significant contributor to the nasal obstruction.
  The Vivaer procedure will be performed in the study clinic using the Vivaer ARC Stylus and Aerin Console. The Vivaer ARC Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device with temperature control capable of delivering very low doses of energy.
  The Vivaer ARC Stylus was cleared for use in the United States (U.S.) by the Food and Drug Administration (FDA) under 510(k) K172529 and the Aerin Console was cleared under 510(k) K162810.
Arm/Group | Single Arm - Vivaer Treatment
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 57
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Nasal Obstruction Symptom Evaluation (NOSE) Scale Mean Change
Description: The primary endpoint is improvement in self-reported Nasal Obstruction Symptom Evaluation (NOSE) Scale score from baseline recorded at the screening evaluation to 13 weeks after the procedure. The NOSE Scale is a validated disease-specific health status instrument used by clinicians to measure the outcome of participants treated for nasal obstruction.43 The NOSE Scale consists of 5 items, each scored using a 5-point Likert scale to make a total score range of 0 through 100, where higher scores indicate worse obstruction. Severity of symptoms can be classified as mild (range, 5-25), moderate (range, 30-50), severe (range, 55-75), or extreme (range, 80-100) nasal obstruction, based on responses to the NOSE Scale survey.
Time Frame: 3 months (13 weeks) visit following screening
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Vivaer Procedure: target population for this study is adults suffering from symptoms attributed to NAO with evidence of SSB obstruction of the airway which may or may not include hypertrophied turbinates. This study requires severe or extreme symptoms demonstrated by a NOSE Scale score ≥ 55 and determination by the investigator that the SSBs are the primary or significant contributor to the nasal obstruction.
Arm/Group | Vivaer Procedure
Number analyzed (Participants) | 69
score on a scale | -45.3 (21.4)

2. Secondary Outcome: Responder Percent
Description: Responder percent: A responder is defined as at least 1 NOSE Scale class improvement or an improvement (decrease) in NOSE Scale score of 20% or more from baseline to 13 weeks after the procedure (eg, going from a score in the severe range (55-75) at preprocedure to a score in the moderate range (30-50) at the 3-month evaluation), or an improvement (decrease) in NOSE Scale score of 20% or more from screening at the 3-month evaluation.
Time Frame: 3 months (13 weeks) visit following baseline
Measure: Number; unit: percentage of responders
Arm/Group | Vivaer Procedure
Number analyzed (Participants) | 69
percentage of responders | 95.7

3. Secondary Outcome: Number of Participants With Device Related Adverse Events
Description: Frequency of device-related and procedure-related serious adverse events, including frequency of septal perforation during the procedure, through the 3-month evaluation.
Time Frame: At or following the study procedure up to 3 months.
Population: AEs with possible relationship to device or procedure. There were no SAEs
Measure: Count of Participants; unit: Participants
Arm/Group | Vivaer Procedure
Number analyzed (Participants) | 69
Participants
  Visual acuity change (transient) | 1
  Nasal scarring at 3M | 2
  Nasal bleeding at 1M | 1
  Nasal Discharge | 2
  Headache | 1
  Nasal Congestion/Obstruction | 1
  Vasovagal reaction | 1
  No Device or Procedure related Issues | 60

ADVERSE EVENTS:
Time Frame: 2 years and 7.5 months
Arm/Group | Vivaer Procedure
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 9/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivaer Procedure (N=69)
Visual Acuity Change (Transient) (Eye disorders) | 1 (1)
Nasal Scarring at 3M (Skin and subcutaneous tissue disorders) | 2 (2)
Nasal Bleeding at 1M (Blood and lymphatic system disorders) | 1 (1)
Nasal Discharge (Skin and subcutaneous tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Nasal Congestion/Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vasovagal Reaction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT05099263/Prot_SAP_000.pdf